CLINICAL TRIAL: NCT04540497
Title: A Phase 3, Randomized, Double-blind, Multicenter, Placebo Controlled Study of Inebilizumab Efficacy and Safety in IgG4-Related Disease
Brief Title: A Study of Inebilizumab Efficacy and Safety in IgG4- Related Disease
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VIB0551.P3.S2; 2023-508290-81-00 (EU CTIS Number)
Expanded Access: NCT06590051 (Available)
Record Dates: First submitted 2020-09-01; First posted 2020-09-07 (Actual); Results first posted 2025-06-25 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: IgG4 Related Disease
MeSH Terms: conditions — Immunoglobulin G4-Related Disease | interventions — inebilizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VIB0551 (Experimental): Inebilizumab administered as an IV infusion.
  Interventions: Drug: Inebilizumab
- Placebo (Placebo Comparator): Placebo administered as an IV infusion.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Inebilizumab — Inebilizumab is a monoclonal antibody that depletes B cells.
  Arms: VIB0551
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study aims to evaluate the efficacy and safety of inebilizumab for the prevention of flare of Immunoglobulin G4-related disease (IgG4-RD).

DETAILED DESCRIPTION:
After a screening period of up to 28 days, subjects with IgG4-RD at high risk of flare due to multi-organ disease and recent active disease will be randomized in a 1:1 ratio to receive intravenous (IV) inebilizumab or placebo after premedication during the 52-week randomized control period (RCP). All subjects will receive an initial tapering dose of glucocorticoids (GCs) to complete treatment of their active disease. Flares occurring during study will be treated. The primary endpoint is time to a first adjudication committee-determined, investigator-treated disease flare during the RCP. The primary analysis will be conducted when the last subject completes the RCP visit or discontinues the RCP. This study includes an optional 3-year open-label treatment period. The study also includes a Safety Follow-up Period (SFUP) of up to 730 days for all participants. The expected duration of each subject's participation in this study is up to 400 days (screening and RCP), plus up to 1095 days for eligible subjects who enroll in the optional open label period (OLP), and up to 730 days for the SFUP, for a total maximum duration of up to 2273 days (screening, RCP, interval between RCP and OLP, OLP, and FSUP).

Study acquired from Horizon in 2024.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female adults, ≥ 18 years of age at time of informed consent.
2. Clinical diagnosis of IgG4-RD.
3. Fulfillment of the 2019 ACR/EULAR classification criteria.
4. Experiencing (or recently experienced) an IgG4-RD flare that requires initiation or continuation of glucocorticoid (GC) treatment at the time of informed consent.
5. IgG4-RD affecting at least 2 organs/sites at any time in the course of IgG4-RD
6. Non-sterilized male subjects who are sexually active with a female partner of childbearing potential must use a condom with spermicide from Day 1 through to the end of the study and must agree to continue using such precautions for at least 6 months after the final dose of IP. Females of childbearing potential who are sexually active with a non-sterilized male partner must use a highly effective method of contraception

Key Exclusion Criteria:

1. History of solid organ or cell-based transplantation or known immunodeficiency disorder.
2. Active malignancy or history of malignancy that was active within the last 10 years (some specific situations for cervical, skin or prostate cancer are acceptable).
3. Receipt of any biologic B cell-depleting therapy or non-depleting B-cell-directed therapy in the 6 months prior to screening.
4. Receipt of non-biologic DMARD or immunosuppressive agent other than GCs within 4 weeks prior to screening.
5. Active tuberculosis or high risk for tuberculosis; hepatitis C infection in absence of curative treatment; evidence of hepatitis B infection.
6. Receipt of live vaccine or live therapeutic infectious agent within 2 weeks prior to screening.
7. Estimated glomerular filtration rate < 30 mL/min/1.73 m^2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2020-12-04 (Actual); Primary Completion 2024-04-09 (Actual); Study Completion 2028-10-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (72):
- United States (4):
  - Viela Bio Investigative Site, Palo Alto, California
  - Viela Bio Investigative Site, Atlanta, Georgia
  - Viela Bio Investigative Site, Baltimore, Maryland
  - Viela Bio Investigative Site, Boston, Massachusetts
- Argentina (2):
  - Viela Bio Investigative Site, Buenos Aires
  - Viela Bio Investigative Site, Mendoza
- Australia (3):
  - Viela Bio Investigative Site, Auchenflower, Queensland
  - Viela Bio Investigative Site, Adelaide, South Australia
  - Viela Bio Investigative Site, Fitzroy
- Canada (3):
  - Viela Bio Investigative Site, Sherbrooke
  - Viela Bio Investigative Site 1, Toronto
  - Viela Bio Investigative Site 2, Toronto
- China (10):
  - Viela Bio Investigative Site, Hohhot, Inner Mongolia
  - Viela Bio Investigative Site 1, Beijing
  - Viela Bio Investigative Site 2, Beijing
  - Viela Bio Investigative Site 3, Beijing
  - Viela Bio Investigative Site 4, Beijing
  - Viela Bio Investigative Site 5, Beijing
  - Viela Bio Investigative Site, Guandong
  - Viela Bio Investigative Site, Shang’ai
  - Viela Bio Investigative Site, Shenyang
  - Viela Bio Investigative Site, Wuhan
- France (5):
  - Viela Bio Investigative Site, Clichy
  - Viela Bio Investigative Site, Lille
  - Viela Bio Investigative Site, Marseille
  - Viela Bio Investigative Site, Nantes
  - Viela Bio Investigative Site, Pessac
- Germany (3):
  - Viela Bio Investigative Site, Berlin
  - Viela Bio Investigative Site, Lübeck
  - Viela Bio Investigative Site, München
- Viela Bio Investigative Site, Hong Kong, Hong Kong
- Hungary (2):
  - Viela Bio Investigative Site, Debrecen
  - Viela Bio Investigative Site, Szeged
- Viela Bio Investigative Site, Bangalore, India
- Viela Bio Investigative Site, Cork, Ireland
- Israel (4):
  - Viela Bio Investigative Site, Kfar Saba
  - Viela Bio Investigative Site, Petah Tikva
  - Viela Bio Investigative Site, Tel Aviv
  - Viela Bio Investigative Site, Tel Litwinsky
- Italy (6):
  - Viela Bio Investigative Site, Florence
  - Viela Bio Investigative Site, Milan
  - Viela Bio Investigative Site, Pisa
  - Viela Bio Investigative Site, Reggio Emilia
  - Viela Bio Investigative Site, Torino
  - Viela Bio Investigative Site, Verona
- Japan (10):
  - Viela Bio Investigative Site, Fukuoka
  - Viela Bio Investigative Site, Hokkaido
  - Viela Bio Investigative Site, Hyōgo
  - Viela Bio Investigative Site, Ishikawa
  - Viela Bio Investigative Site, Kyoto
  - Viela Bio Investigative Site, Niigata
  - Viela Bio Investigative Site 2, Osaka
  - Viela Bio Investigative Site, Osaka
  - Viela Bio Investigative Site, Tokyo
  - Viela Bio Investigative Site, Toyama
- Viela Bio Investigative Siite, Tlalpan, Mexico
- Netherlands (2):
  - Viela Bio Investigative Site, Amsterdam
  - Viela Bio Investigative Site, Rotterdam
- Poland (2):
  - Viela Bio Investigative Site, Warsaw
  - Viela Bio Investigative Site, Wroclaw
- Spain (4):
  - Viela Bio Investigative Site 2, Barcelona
  - Viela Bio Investigative Site, Barcelona
  - Viela Bio Investigative Site, Madrid
  - Viela Bio Investigative Site, Valencia
- Sweden (2):
  - Viela Bio Investigative Site, Gothenburg
  - Viela Bio Investigative Site, Stockholm
- Turkey (Türkiye) (2):
  - Viela Bio Investigative Site, Ankara
  - Viela Bio Investigative Site, Istanbul
- United Kingdom (4):
  - Viela Bio Investigative Site, Leeds
  - Viela Bio Investigative Site, London
  - Viela Bio Investigative Site, Newcastle
  - Viela Bio Investigative Site, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stone JH, Khosroshahi A, Zhang W, Della Torre E, Okazaki K, Tanaka Y, Lohr JM, Schleinitz N, Dong L, Umehara H, Lanzillotta M, Wallace ZS, Ebbo M, Webster GJ, Martinez Valle F, Nayar MK, Perugino CA, Rebours V, Dong X, Wu Y, Li Q, Rampal N, Cimbora D, Culver EL; MITIGATE Trial Investigators. Inebilizumab for Treatment of IgG4-Related Disease. N Engl J Med. 2025 Mar 27;392(12):1168-1177. doi: 10.1056/NEJMoa2409712. Epub 2024 Nov 14. PMID 39541094
- [Derived] Perugino C, Culver EL, Khosroshahi A, Zhang W, Della-Torre E, Okazaki K, Tanaka Y, Lohr M, Schleinitz N, Falloon J, She D, Cimbora D, Stone JH. Efficacy and Safety of Inebilizumab in IgG4-Related Disease: Protocol for a Randomized Controlled Trial. Rheumatol Ther. 2023 Dec;10(6):1795-1808. doi: 10.1007/s40744-023-00593-7. Epub 2023 Oct 4. PMID 37792260

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants affected by immunoglobulin G4-related disease (IgG4-RD) were recruited across 46 sites in Argentina, Australia, Canada, China, France, Germany, Israel, Italy, Japan, Mexico, Netherlands, Poland, Spain, Turkey, the United Kingdom and the United States, between December 2020 and February 2024 which was the safety data cutoff date.
Pre-assignment Details: After a 28-day screening period, participants entered a 52-week randomized controlled period (RCP), followed by an optional 3-year open-label period (OLP). The study also included a 2-year safety follow-up (SFUP). The study is ongoing; efficacy data covers the 52-week RCP, while safety data, including 90 participants, were collected up to the cut-off date in February 2024.
Groups:
- RCP: Placebo/OLP: Inebilizumab 300 mg: Participants with IgG4-RD were randomized to receive placebo intravenous (IV) infusion on Day 1, Day 15, and Week 26 during the 52-week RCP. Treatment assignment was stratified based on whether the participant was newly diagnosed or had a recurrent IgG4-RD manifestation. After completing the RCP, participants had the option to enter the optional 3-year OLP, where they received inebilizumab on OLP Days 1 and 15. Participants then received inebilizumab every 6 months (Q6M) for the duration of the OLP.
- RCP: Inebilizumab 300 mg/OLP: Inebilizumab 300 mg: Participants with IgG4-RD were randomized to receive inebilizumab 300 mg IV infusion on Day 1, Day 15, and Week 26 during the 52-week RCP. Treatment assignment was stratified based on whether the participant was newly diagnosed or had a recurrent IgG4-RD manifestation. After completing the RCP, participants had the option to enter the optional 3-year OLP, where they received inebilizumab on OLP Day 1 and matching placebo on Day 15. Participants then received inebilizumab Q6M for the duration of the OLP.
Period: Overall Study
Arm/Group | RCP: Placebo/OLP: Inebilizumab 300 mg | RCP: Inebilizumab 300 mg/OLP: Inebilizumab 300 mg
Started | 67 | 68
Started Optional OLP | 49 | 53
Completed (Participants who completed the 52-week RCP) | 63 | 64
Not Completed | 4 | 4
Not completed — Adverse Event | 0 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Miscellaneous | 2 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: all participants who received any dose of investigational product during the RCP.
Groups:
- Placebo: Participants with IgG4-RD were randomized to receive placebo IV infusion on Day 1, Day 15, and Week 26 during the 52-week RCP. Treatment assignment was stratified based on whether the participant was newly diagnosed or had a recurrent IgG4-RD manifestation. After completing the RCP, participants had the option to enter the optional 3-year OLP, where they received inebilizumab on OLP Days 1 and 15. Participants then received inebilizumab every 6 months (Q6M) for the duration of the OLP.
- Inebilizumab 300 mg: Participants with IgG4-RD were randomized to receive inebilizumab 300 mg IV infusion on Day 1, Day 15, and Week 26 during the 52-week RCP. Treatment assignment was stratified based on whether the participant was newly diagnosed or had a recurrent IgG4-RD manifestation.
- Total: Total of all reporting groups
Arm/Group | Placebo | Inebilizumab 300 mg | Total
Number analyzed (Participants) | 67 | 68 | 135
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.2 (12.2) | 58.2 (11.5) | 58.2 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 29 | 47
  Male | 49 | 39 | 88
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 8 | 16
  Not Hispanic or Latino | 53 | 56 | 109
  Unknown or Not Reported | 6 | 4 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 25 | 38 | 63
  Black or African American | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  White | 32 | 21 | 53
  Other | 2 | 2 | 4
  Unknown | 1 | 0 | 1
  Not Reported | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: RCP: Time to Disease Flare
Description: Time to disease flare was defined as the number of days from Day 1 (dosing) to the date of the first treated and Adjudication Committee (AC)-determined IgG4-RD flare within the 52-week RCP. The date of disease flare was determined by the initiation of any flare treatment, including new or increased glucocorticoid (GC) treatment, other immunotherapy, or an interventional procedure, as deemed necessary by the Investigator to address the flare.
  Kaplan-Meier (KM) method was used to estimate the median time to flare, and 95% confidence interval (CI).
Time Frame: Up to Week 52
Population: Full Analysis Set: all participants who received any dose of investigational product during the RCP.
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Placebo: Participants with IgG4-RD were randomized to receive placebo IV infusion on Day 1, Day 15, and Week 26 during the 52-week RCP. Treatment assignment was stratified based on whether the participant was newly diagnosed or had a recurrent IgG4-RD manifestation.
Arm/Group | Placebo | Inebilizumab 300 mg
Number analyzed (Participants) | 67 | 68
Days | 246.0 [191.0 to NA] — Due to the low level of events of disease flare, the upper limit of the CI could not be calculated using the KM method. | NA [371.0 to NA] — Due to the low level of events of disease flare, the median time to disease flare, and the upper limit of the CI could not be calculated using the KM method.
Statistical Analysis 1: Comparison: Placebo vs Inebilizumab 300 mg; Test type: Other; Hazard Ratio (HR) = 0.13, 95% CI 2-sided [0.06 to 0.28] — Inebilizumab versus placebo

2. Secondary Outcome: RCP: Annualized Rate of Treated and AC-Determined Flares During the RCP
Description: The annualized rate of treated and AC-determined flares during the 52-week RCP was calculated by dividing the total number of treated and AC-determined flares by the total time at risk (in years) for all participants. This measure reflected the frequency of disease flares per person per year during the RCP.
Time Frame: Week 52
Population: Full Analysis Set: all participants who received any dose of investigational product during the RCP.
Measure: Number (95% Confidence Interval); unit: Flares per person per year
Arm/Group | Placebo | Inebilizumab 300 mg
Number analyzed (Participants) | 67 | 68
Flares per person per year | 0.71 [0.53 to 0.94] | 0.10 [0.05 to 0.21]

3. Secondary Outcome: RCP: Percentage of Participants Achieving Flare-free, Treatment-free Complete Remission at Week 52
Description: Flare-free, treatment-free complete remission at Week 52 was defined as the absence of evident disease activity at Week 52, no AC-determined flare during the RCP, and no treatment for flare or disease control, except for the required 8-week glucocorticoid taper. Lack of evident disease activity was determined by either a score of 0 on the IgG4-RD Responder Index (score range: 0-4, with lower scores indicating better disease control) or an investigator's assessment that no disease activity was present based on physical, laboratory, pathology, or other evidence.
Time Frame: Week 52
Population: Full Analysis Set: all participants who received any dose of investigational product during the RCP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Inebilizumab 300 mg
Number analyzed (Participants) | 67 | 68
Participants | 15 | 39

4. Secondary Outcome: RCP: Percentage of Participants Achieving Flare-free, Corticosteroid-free Complete Remission at Week 52
Description: Flare-free, corticosteroid-free complete remission at Week 52 was defined as the absence of evident disease activity at Week 52, no AC-determined flare during the RCP, and no corticosteroid treatment for flare or disease control, except for the required 8-week glucocorticoid taper. Lack of evident disease activity was determined by either a score of 0 on the IgG4-RD Responder Index (score range: 0-4, with lower scores indicating better disease control) or an investigator's assessment that no disease activity was present based on physical, laboratory, pathology, or other evidence.
Time Frame: Week 52
Population: Full Analysis Set: all participants who received any dose of investigational product during the RCP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Inebilizumab 300 mg
Number analyzed (Participants) | 67 | 68
Participants | 15 | 40

5. Secondary Outcome: Number of Participants Who Experienced Treatment-emergent Adverse Events (TEAEs) During the RCP
Description: An adverse event (AE) referred to any untoward medical occurrence in a clinical study participant, regardless of a causal relationship with the study treatment. TEAEs included any event occurring after the participant received the study treatment. Clinically significant changes in vital signs, electrocardiograms, and laboratory tests recorded after treatment administration were documented as TEAEs. Serious AEs (SAEs) were untoward medical occurrences after the first dose, irrespective of a causal link to the study treatment, that led to death, were life-threatening, required hospitalization or its prolongation, caused significant disability, resulted in congenital anomalies, or were considered other medically important events. AEs were graded (Grade 3: severe; Grade 4: life-threatening; Grade 5: death) using the Common Terminology Criteria for Adverse Events [CTCAE]).
Time Frame: Up to Week 52
Population: Safety Analysis Set RCP: All participants who received any dose of investigational product during the RCP. Participants were analyzed according to the treatment they actually received. Specifically, participants randomized to the inebilizumab group who received all placebo dose were included in the placebo group.
Measure: Count of Participants; unit: Participants
Groups:
- Inebilizumab 300 mg: Participants with IgG4-RD were randomized to receive inebilizumab 300 mg IV infusion on Day 1, Day 15, and Week 26 during the 52-week RCP. Treatment assignment was stratified based on whether the participant was newly diagnosed or had a recurrent IgG4-RD manifestation. After completing the RCP, participants had the option to enter the optional 3-year OLP, where they received inebilizumab on OLP Day 1 and matching placebo on Day 15. Participants then received inebilizumab Q6M for the duration of the OLP.
Arm/Group | Placebo | Inebilizumab 300 mg
Number analyzed (Participants) | 67 | 68
Participants
  TEAEs | 66 | 66
  SAEs | 6 | 12
  Fatal TEAEs | 0 | 0
  Grade ≥ 3 TEAEs | 8 | 12

6. Secondary Outcome: Number of Participants Who Experienced TEAEs During the OLP
Description: An AE referred to any untoward medical occurrence in a clinical study participant, regardless of a causal relationship with the study treatment. TEAEs included any event occurring after the participant received the study treatment. Clinically significant changes in vital signs, electrocardiograms, and laboratory tests recorded after treatment administration were documented as TEAEs. SAEs were untoward medical occurrences after the first dose, irrespective of a causal link to the study treatment, that led to death, were life-threatening, required hospitalization or its prolongation, caused significant disability, resulted in congenital anomalies, or were considered other medically important events. AEs were graded (Grade 3: severe; Grade 4: life-threatening; Grade 5: death) using the CTCAE).
Time Frame: From the first dose of investigational product in OLP to the end of OLP or cutoff date; median (min, max) duration was 51.6 (0.1, 108.3) weeks.
Reporting Status: Not Posted, anticipated posting 2029-10

7. Secondary Outcome: RCP: Number of Participants With Anti-drug Antibodies (ADA) to Inebilizumab by Week 52
Description: Incidence was the proportion of the participants with ADA positive post-baseline only or boosted their preexisting ADA (at least 4-fold over the baseline titer) during the study period. Baseline was defined as the last valid value on or before the first dose of RCP.
Time Frame: Baseline to Week 52
Population: Full Analysis Set: all participants who received any dose of investigational product during the RCP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Inebilizumab 300 mg
Number analyzed (Participants) | 67 | 68
Participants | 5 | 6

8. Secondary Outcome: RCP: Time to Initiation of First Treatment for New or Worsening Disease Activity Within the RCP
Description: Time to initiation of the first treatment (medication or procedure) for new or worsening disease activity, as determined by the investigator, within the RCP, was measured from day 1 (dosing) to the date the first treatment was administered. It Included any treatment initiated by the investigator for disease activity, regardless of the AC determination of flare.
  KM method was used to estimate the median time to the initiation of first treatment or worsening of disease activity, and 95% CI.
Time Frame: Week 52
Population: Full Analysis Set: all participants who received any dose of investigational product during the RCP, and experienced IgG4-RD flares, regardless of the AC determination of flare.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo | Inebilizumab 300 mg
Number analyzed (Participants) | 42 | 7
Days | 237.0 [143.0 to 310.0] | NA [371.0 to NA] — Due to insufficient number of participants initiating a new treatment or worsening disease activity, the median and upper CI were not reached using the KM method.
Statistical Analysis 1: Comparison: Placebo vs Inebilizumab 300 mg; Test type: Other; Hazard Ratio (HR) = 0.12, 95% CI 2-sided [0.05 to 0.26] — Inebilizumab vs placebo

9. Secondary Outcome: RCP: Annualized Flare Rate for AC-Determined IgG4-RD Flares at Week 52
Description: The annualized flare rate for AC-determined IgG4-RD flares, whether or not treated, during the RCP was calculated by dividing the total number of AC-determined flares by the total time at risk (in years) for all participants. This measure reflected the frequency of IgG4-RD flares, irrespective of treatment, per participant per year during the study period.
Time Frame: Week 52
Population: Full Analysis Set: all participants who received any dose of investigational product during the RCP.
Measure: Number (95% Confidence Interval); unit: Flares per participant per year
Arm/Group | Placebo | Inebilizumab 300 mg
Number analyzed (Participants) | 67 | 68
Flares per participant per year | 0.75 [0.57 to 0.99] | 0.16 [0.09 to 0.29]

10. Secondary Outcome: RCP: Cumulative Glucocorticoid (GC) Use for IgG4-RD Disease Control by Week 52
Description: GC use was calculated as the cumulative glucocorticoid dose (in milligrams) taken for the purpose of IgG4-RD disease control during the RCP. This measure accounted for all GC treatments administered to participants to manage disease activity throughout the study period.
Time Frame: Week 52
Population: Full Analysis Set: all participants who received any dose of investigational product during the RCP.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Placebo | Inebilizumab 300 mg
Number analyzed (Participants) | 67 | 68
mg | 1384.53 (1723.26) | 118.25 (438.97)

ADVERSE EVENTS:
Time Frame: For RCP mortality reporting: from randomization to the end of RCP; median (min, max) was 54.1 (2.1, 65.1) weeks. For RCP AE reporting: from Day 1 to the end of RCP or cutoff date; median (min, max) was 54.1 (2.1, 65.1) weeks. For OLP mortality and AE reporting: from the 1st dose of IP in OLP to the end of OLP or cutoff date; median (min, max) was 51.6 (0.1, 108.3) weeks.
Description: Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug. All-cause mortality is reported for all participants randomized in the study.
Groups:
- RCP: Placebo: Participants with IgG4-RD were randomized to receive placebo IV infusion on Day 1, Day 15, and Week 26 during the 52-week RCP. Treatment assignment was stratified based on whether the participant was newly diagnosed or had a recurrent IgG4-RD manifestation.
- RCP: Inebilizumab 300 mg: Participants with IgG4-RD were randomized to receive inebilizumab 300 mg IV infusion on Day 1, Day 15, and Week 26 during the 52-week RCP.
- OLP: Inebilizumab 300 mg: Participants received inebilizumab on OLP Days 1 and 15. Participants then received inebilizumab Q6M for the duration of the OLP.
Arm/Group | RCP: Placebo | RCP: Inebilizumab 300 mg | OLP: Inebilizumab 300 mg
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/68 | 0/90
Serious Adverse Events (participants affected / at risk) | 6/67 | 12/68 | 14/90
Other Adverse Events (participants affected / at risk) | 49/67 | 54/68 | 51/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RCP: Placebo (N=67) | RCP: Inebilizumab 300 mg (N=68) | OLP: Inebilizumab 300 mg (N=90)
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 1 | 1
Dengue fever (Infections and infestations) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Febrile infection (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Fibroadenomatoid mastopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary atypical adenomatous hyperplasia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lichen sclerosus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RCP: Placebo (N=67) | RCP: Inebilizumab 300 mg (N=68) | OLP: Inebilizumab 300 mg (N=90)
Lymphopenia (Blood and lymphatic system disorders) | 6 | 11 | 1
Neutropenia (Blood and lymphatic system disorders) | 3 | 4 | 3
Palpitations (Cardiac disorders) | 1 | 4 | 1
Abdominal pain (Gastrointestinal disorders) | 7 | 4 | 3
Abdominal pain upper (Gastrointestinal disorders) | 5 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 9 | 3 | 2
Nausea (Gastrointestinal disorders) | 4 | 0 | 1
Asthenia (General disorders) | 8 | 2 | 1
Fatigue (General disorders) | 5 | 5 | 4
Pyrexia (General disorders) | 3 | 6 | 4
COVID-19 (Infections and infestations) | 13 | 15 | 19
Conjunctivitis (Infections and infestations) | 4 | 1 | 2
Nasopharyngitis (Infections and infestations) | 4 | 6 | 5
Sinusitis (Infections and infestations) | 4 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 8 | 4 | 10
Urinary tract infection (Infections and infestations) | 4 | 8 | 3
Alanine aminotransferase increased (Investigations) | 4 | 2 | 1
Gamma-glutamyltransferase increased (Investigations) | 3 | 4 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 4 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 6 | 3
Immunoglobulin G4 related disease (Musculoskeletal and connective tissue disorders) | 5 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 4 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 2 | 0
Dizziness (Nervous system disorders) | 5 | 1 | 1
Headache (Nervous system disorders) | 7 | 6 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 3
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 3 | 1
Hypertension (Vascular disorders) | 2 | 1 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2023-08-08): https://cdn.clinicaltrials.gov/large-docs/97/NCT04540497/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-15): https://cdn.clinicaltrials.gov/large-docs/97/NCT04540497/SAP_001.pdf